CLINICAL TRIAL: NCT03398122
Title: Study of Apatinib Combined With TACE in Advance Hepatocellular Carcinoma
Acronym: HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-HBH001
Record Dates: First submitted 2018-01-07; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Apatinib; advanced hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib combined with TACE (Experimental): patients received Aptinib, 250 mg daily after TACE treatment, for 4-6 weeks
  Interventions: Procedure: TACE; Drug: Apatinib
- chemoemtranscatherer arterial bolization (Placebo Comparator): epirubicin 30-60mg was injected into the blood supply artery of the tumor ,Embolization was subsequently performed with granules of gelatin sponge particles.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Procedure: TACE — epirubicin 30-60mg was injected into the blood supply artery of the tumor ,Embolization was subsequently performed with granules of gelatin sponge particles.
  Other Names: chemoemtranscatherer arterial bolization
  Arms: Apatinib combined with TACE
Drug: Apatinib — a molecular targeted anti-tumor drugs,small molecule vascular endothelial growth factor receptor 2 inhibitor
  Other Names: ai tan

SUMMARY:
the purpose of this study is to evaluate the efficacy and safety of aptinib in patients with advanced HCC

DETAILED DESCRIPTION:
HCC The is a common malignancy in the world, especially in China. Advanced HCC treatment is difficult and the prognosis is poor, which is still a great challenge and threat to the medical profession. The advent of the molecular targeted drug, Sola, has made the treatment dilemma of advanced HCC a breakthrough, but the efficacy and economic health ratio is far from satisfactory. After Sola, many new molecular targeted drugs were studied, but failed.

Although multiple treatment options, but for HCC Patient-recommended treatment programs require systematic treatment and surgery, TACE , local ablation and radiotherapy and other multidisciplinary means of combination, the selection of appropriate patients, appropriate means and timing to achieve individualized treatment.

1. Aptinib Union TACE can be generated through embolization and angiogenesis by the dual target of vascular suppression;2. TACE induces hypoxia, leading to an increase in the number of hypoxia-inducing factors that increases VEGF and PDGFR , while VEGF the and PDGFR may be important factors that induce tumor recurrence by stimulating tumor angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old;
2. initial treatment diagnosed by histopathological or cytological examination BCLC Staging B/C Hepatocellular carcinoma of the liver ( HCC ) and at least one of the largest tumors in measurable lesions ≤15cm ;
3. Child-pugh liver function Rating: A level, B level;
4. BCLC Staging as B / C period;
5. before join in the group 1 weeks ECOG PS Rating: 0-1 score; estimated Lifetime ≥12 Week; Lab metrics meet the following criteria: ( 1 ) Blood routine check:

   1. HB≥90 g/L;
   2. ANC≥1.5x109/L;
   3. PLT≥60x109/L; ( 2 ) Biochemical Examination:

   <!-- -->

   1. ALB≥29 g/L;
   2. ALT and AST<2.5*ULN;
   3. TBIL ≤ 2*ULN;
   4. Cr ≤ 1.5*ULN;
6. women of childbearing age must be pregnancy tests before join in the group in 7 days;
7. Participants volunteered to join this study should sign informed consent, with good compliance and follow-up.

Exclusion Criteria:

1. Central hepatic artery / hepatic venous fistula in patients with hepatocellular carcinoma, diffuse liver cancer patients, with large vascular invasion of liver cancer patients (including portal vein tumor thrombus);
2. hepatobiliary cell carcinoma and mixed cell carcinoma are known; previous ( 5 year) or at the same time suffering from other incurable malignancies, except for the cured basal cell carcinoma of the skin and cervical carcinoma in situ;
3. clinically symptomatic ascites that requires therapeutic celiac puncture or drainage with high blood pressure and cannot be reduced to normal range by anti hypertensive medications (systolic pressure > 140 mmHg , diastolic pressure >90 mmHg );
4. Suffering Ⅱ above-level myocardial ischemia or myocardial infarction, control of poor arrhythmia (including QTC inter-phase male ≥450 ms , female ≥470 ms );
5. Follow NYHA Standard Ⅲ ~ Ⅳ grade heart insufficiency or heart color Doppler ultrasonography: LVEF (left ventricular ejection fraction) < 50% ;
6. There are various factors affecting oral medication (e.g.inability to swallow, chronic diarrhea and intestinal obstruction, which significantly affect drug use and absorption);
7. previous within 6 months there is a history of gastrointestinal bleeding or a clear tendency to gastrointestinal bleeding, such as: bleeding risk of esophageal varices, local active ulcer lesions, fecal occult blood ≥ ( ++ ) not in group; fecal occult blood (+ ), requiring gastroscopy;
8. before participating in this study There were abdominal fistula, gastrointestinal perforation or celiac abscess in the day;
9. Coagulation dysfunction ( INR > 1.5 or prothrombin time ( PT ) > ULN+4 seconds), with bleeding tendencies or undergoing thrombolysis or anticoagulant therapy;
10. patients who have undergone central nervous system metastasis or known brain metastases;
11. patients with objective evidence of the history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, and severe lung impairment;
12. urine proteins are routinely shown ≥++ or confirmed 24 hour urine protein ration > 1.0 g ;
13. before participating in the study 7 days use strong-effect in CYP3A4 inhibitor therapy, or prior to participating in the study 12 days use the strong-effect in CYP3A4 inducer Therapy;
14. pregnant or lactating women who are not willing or unable to take effective contraceptive measures;
15. A history of mental illness, or psychotropic substance abuse;
16. Union HIV infected patients;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
PFS | one and a half year
  progression free survival

SECONDARY OUTCOMES:
OS | one and a half year
  overall survival
TTP | one and a half year
  time to progression
DCR | one and a half year
  disease control rate
ORR | one and a half year
  objective response rate
QOL | one and a half year
  number of participants with treatment-related adverse events as assessed by EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Guo, MD, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China